CLINICAL TRIAL: NCT01244893
Title: Study of ACUVUE® ADVANCE® PLUS Contact Lenses.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-1636BI
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Results first posted 2014-02-03 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2017-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Acuvue Advance Plus prePQ/Acuvue Advance Plus postPQ (Other): Acuvue Advance Plus silicone hydrogel contact lens manufactured prior to process qualification will be worn first and Acuvue AdvancePlus silicone hydrogel contact lens manufactured after process qualification will be worn second.
  Interventions: Device: Acuvue Advance Plus prePQ; Device: Acuvue Advance Plus postPQ
- Acuvue Advance Plus postPQ/Acuvue Advance Plus prePQ (Other): Acuvue Advance Plus silicone hydrogel contact lens manufactured prior to process qualification worn first and Acuvue Advance Plus silicone hydrogel contact lens manufactured after process qualification worn second.
  Interventions: Device: Acuvue Advance Plus prePQ; Device: Acuvue Advance Plus postPQ

INTERVENTIONS:
Device: Acuvue Advance Plus prePQ — silicone hydrogel contact lens manufactured prior to equipment process qualification activities.
Device: Acuvue Advance Plus postPQ — silicone hydrogel contact lens manufactured after equipment process qualification activities.

SUMMARY:
The purpose of this study is to compare ACUVUE® ADVANCE® Plus contact lenses made prior to process qualification (prePQ) against the ACUVUE® ADVANCE® Plus lenses made after the process qualification (postPQ).

ELIGIBILITY:
Inclusion Criteria:

* The subject must be at least 18 years of age and no more than 39 years of age.
* The subject is a current spherical soft contact lens wearer and willing to wear the study lenses on a daily wear basis for the duration of the study (minimum of 6 hours per day).
* The subject's optimal vertexed spherical equivalent distance correction must be between -1.00 and - 5.00D.
* Any cylinder power must be ≤ -0.75D.
* The subject must have visual acuity best correctable to 20/25+3 or better for each eye.
* The subject must read and sign the Statement of Informed Consent.
* The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.

Exclusion Criteria:

* Ocular or systemic allergies or disease which might interfere with contact lens wear.
* Systemic disease or use of medication which might interfere with contact lens wear.
* Clinically significant (grade 3 or 4) corneal edema, corneal vascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear.
* Clinically significant (grade 3 or 4) tarsal abnormalities or bulbar injection which might interfere with contact lens wear.
* Any ocular infection.
* Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
* Pregnancy or lactation.
* Diabetes.
* Infectious diseases (e.g. hepatitis, tuberculosis) or an immuno-suppressive disease (e.g. HIV).
* Habitual contact lens type is toric, multifocal, or is worn as extended wear.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Powell, Ohio
  - Warwick, Rhode Island
  - Salem, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4 investigation sites were used within the U.S. for this study, with a study duration of Oct 23, 2010 to Nov 7, 2010.
Pre-assignment Details: 44 subjects enrolled; 42 completed as cohort, two subjects were discontinued.
Groups:
- Acuvue Advance Plus preQ/Acuvue Advance Plus postQ: Arm 1:
  Acuvue Advance Plus silicone hydrogel contact lens manufactured prior to qualification were worn first, then Acuvue AdvancePlus silicone hydrogel contact lens manufactured after qualification were worn second.
  Arm 2:
  Acuvue AdvancePlus silicone hydrogel contact lens manufactured after qualification were worn first, then Acuvue Advance Plus silicone hydrogel contact lens manufactured prior to qualification were worn second.
- Acuvue Advance Plus postQ/Acuvue Advance Plus preQ: Arm 1:
  Acuvue Advance Plus silicone hydrogel contact lens manufactured prior to qualification will be worn first, then Acuvue AdvancePlus silicone hydrogel contact lens manufactured after qualification will be worn second.
  Arm 2:
  Acuvue AdvancePlus silicone hydrogel contact lens manufactured after qualification will be worn first, then Acuvue Advance Plus silicone hydrogel contact lens manufactured prior to qualification will be worn second.
Period: Baseline
Arm/Group | Acuvue Advance Plus preQ/Acuvue Advance Plus postQ | Acuvue Advance Plus postQ/Acuvue Advance Plus preQ
Started | 22 | 22
Completed | 22 | 21
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1
Period: 1-Week Follow Up
Arm/Group | Acuvue Advance Plus preQ/Acuvue Advance Plus postQ | Acuvue Advance Plus postQ/Acuvue Advance Plus preQ
Started | 22 | 21
Completed | 21 | 21
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Final Visit
Arm/Group | Acuvue Advance Plus preQ/Acuvue Advance Plus postQ | Acuvue Advance Plus postQ/Acuvue Advance Plus preQ
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 44 persons enrolled, 42 completed as cohort, 2 dropped due to: 1 non-trial related adverse event, and 1 protocol deviation
Groups:
- All Subjects: Acuvue Advance Plus silicone hydrogel contact lens manufactured prior to qualification were worn first and Acuvue AdvancePlus silicone hydrogel contact lens manufactured after qualification were worn second.
Arm/Group | All Subjects
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (5.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity (VA)
Description: Snellen VA was measured to the nearest letter then converted to the logMAR scale for the analysis. Values < 0 imply a clinically positive result; while values > 0 infer a clinically negative result.
Time Frame: 6-8 days after lens wear
Population: Population analyzed are those who were enrolled, randomized, and completed the study.
Measure: Mean (Standard Deviation); unit: logMAR scale
Groups:
- Acuvue Advance Plus preQ: Acuvue Advance Plus silicone hydrogel contact lens manufactured prior to qualification were worn daily for 6-8 days. Binocular measurements reported only.
- Acuvue Advance Plus postQ: Acuvue Advance Plus silicone hydrogel contact lens manufactured post qualification were worn daily for 6-8 days. Binocular measurements reported only.
Arm/Group | Acuvue Advance Plus preQ | Acuvue Advance Plus postQ
Number analyzed (Participants) | 42 | 42
logMAR scale | -0.088 (0.0328) | -0.083 (0.0377)
Statistical Analysis 1: Comparison: Acuvue Advance Plus preQ vs Acuvue Advance Plus postQ; Ho: after time period (6-8 days of lens wear), the test lens - control lens will be greater than or equal to the non-inferiority margin specified . Ha: after time period, test-control will be less than the margin specified concluding that the test lens will be inferior to control lens in terms of LogMAR scale; Test type: Non-Inferiority or Equivalence — This study uses -0.05 LogMAR as the non-inferiority margin; Mixed Models Analysis; Mean Difference (Final Values) = 0.005, 95% CI 2-sided [-0.00092 to 0.01045], Standard Error of Mean 0.003 — The mean difference is calculated as the test lens - control lens

2. Secondary Outcome: Corneal Staining
Description: Corneal staining type was assessed by Investigator using a slit lamp and graded on a 5-point scale; 0=none, 1=trace, 2=mild, 3=moderate, 4=severe.
Time Frame: 6-8 days after lens wear
Population: Population analyzed are those who were enrolled, randomized, and completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Groups:
- Acuvue Advance Plus preQ: Acuvue Advance Plus silicone hydrogel contact lens manufactured prior to qualification were worn daily for 6-8 days.
- Acuvue Advance Plus postQ: Acuvue Advance Plus silicone hydrogel contact lens manufactured post to qualification were worn daily for 6-8 days.
Arm/Group | Acuvue Advance Plus preQ | Acuvue Advance Plus postQ
Number analyzed (Participants) | 42 | 42
Number analyzed (eyes) | 74 | 78
units on a scale | 0.23 (0.424) | 0.17 (0.375)

3. Secondary Outcome: Limbal Redness
Description: Limbal redness was assessed by using a 5-point scale: 0=none, 1=trace, 2=mild, 3=moderate, 4=severe.
Time Frame: 6-8 days after lens wear
Population: Population analyzed are those who were enrolled, randomized, and completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Acuvue Advance Plus postQ: Acuvue Advance Plus silicone hydrogel contact lens manufactured post qualification were worn daily for 6-8 days.
Arm/Group | Acuvue Advance Plus preQ | Acuvue Advance Plus postQ
Number analyzed (Participants) | 42 | 42
units on a scale | 0.71 (0.457) | 0.79 (0.682)

4. Secondary Outcome: Bulbar Redness
Description: Scale of 0 increasing to 4. 0=None, 4=Severe Redness
Time Frame: 6-8 days after lens wear
Population: Population analyzed consisted of those who were enrolled, randomized, and completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Acuvue Advance Plus preQ: Acuvue Advance Plus silicone hydrogel contact lens manufactured prior to qualification were worn daily for 6-9 days.
- Acuvue Advance Plus postQ: Acuvue Advance Plus silicone hydrogel contact lens manufactured post qualification were worn daily for 6-9 days.
Arm/Group | Acuvue Advance Plus preQ | Acuvue Advance Plus postQ
Number analyzed (Participants) | 42 | 42
units on a scale | 0.71 (0.673) | 0.71 (0.596)

ADVERSE EVENTS:
Groups:
- AAP PreQ; AAP PostQ: Acuvue Advance Plus silicone hydrogel contact lenses will be used both pre- / post-qualification.
Arm/Group | AAP PreQ | AAP PostQ
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No